CLINICAL TRIAL: NCT00888342
Title: A Study of Changes in Blood Gases, Disturbance of Breath During Sleep and Cardiovascular Co-morbidity in Patients With COPD in Different Stages of the Disease, and the Effect of Alcohol, Supplementary Oxygen and Zopiclone on These Changes.
Brief Title: Changes in Blood Gases, Disturbance of Breath During Sleep and Cardiovascular Co-morbidity in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); Landsforeningen for hjerte og lungesyke (LHL) (Unknown); University Hospital, Akershus (Other); Haukeland University Hospital (Other); ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GK-61; 2008/2/0083 (LHL) (Other Grant/Funding Number: Landsforeningen for Hjerte og Lungesyke (LHL)); 2688 (BIOBANK) (Registry Identifier: The National Committees for Research Ethics in Norway); 6.2009.10 (REK) (Registry Identifier: The National Committees for Research Ethics in Norway)
Record Dates: First submitted 2009-04-22; First posted 2009-04-27 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Disease; Chronic Obstructive; Hypercapnia; Hypoxemia; Arrhythmias, Cardiac
Keywords: Pulmonary Disease; Chronic Obstructive; Hypercapnia; Hypoxemia; Arrhythmias, Cardiac; Polysomnography; Capnography; Electrocardiography, Holter
MeSH Terms: conditions — Lung Diseases; Hypercapnia; Hypoxia; Arrhythmias, Cardiac | interventions — zopiclone; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 supplementary oxygen (Active Comparator): participant receives supplementary oxygen one night, polysomnography with capnography will be compared to no treatment another night
  Interventions: Drug: supplementary oxygen
- 2 Zopiclone (Active Comparator): participant receives 5 mg zopiclone one night, polysomnography with capnography will be compared to no treatment another night
  Interventions: Drug: zopiclone
- 3 Alcohol (Active Comparator): participant receives 0,5 mg alcohol /kg body weight before sleep one night, polysomnography with capnography will be compared to no intervention another night
  Interventions: Other: alcohol

INTERVENTIONS:
Drug: supplementary oxygen — Supplementary oxygen 2 L/min if SpO2 < 90%. If SpO2 < 90 % the oxygen dose is titrated until SpO2 reads 88-92%. For patients on LTOT the oxygen dose is doubled for intervention.
  Other Names: 100% oxygen gas with continous flow from wall outlet
  Arms: 1 supplementary oxygen
Drug: zopiclone — 5 mg sedative given approximately 1 hour before sleep
  Other Names: Imovane, Zopiklon
  Arms: 2 Zopiclone
Other: alcohol — 5 mg alcohol/kg body-weight approximately 1 hour before sleep
  Other Names: 96% ethanol
  Arms: 3 Alcohol

SUMMARY:
Respiration failure type 2 is loss of the lungs ability to take up oxygen (O2) and get rid of carbon dioxide (CO2). The diagnosis is based on blood gas measurement of pressures of O2 and CO2. Patients with COPD is often seen to have co-morbidity with cardiac diseases. Chronic systemic inflammation is seen in both COPD and cardiac diseases. The investigators will investigate the sleep quality, CO2-retention, O2-saturation, cardiac arrythmias and markers of inflammation in 120 patients with COPD in different stages of the disease. Our hypotheses are:

* that the first signs of respiration failure type 2 is seen during sleep with alteration of sleep patterns and greater and more long-lasting retention of CO2 in the blood compared to those with a normal lung function
* that the use of alcohol, zopiclone or supplementary oxygen will make these differences even greater
* that cardiac arrythmias correlates with hypoxemia
* that cardiac arrythmias and respiration failure correlates with degree of inflammation

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1 < 80 % of pred. and FEV1/FVC < 0,7)

Exclusion Criteria:

* other serious disease (like lung cancer, sarcoidosis, restrictive lung disease)
* exacerbation of COPD within 3 weeks before inclusion
* coronary heart disease with unstable angina pectoris or myocardial infarction within 3 months of incl.
* uncontrolled hypertension
* cerebral infarction
* neurological, muscular or skeletal disease/disorder that affect abdominal- and/or thoracal movements (kyphoscoliosis, paresis, etc)
* unstable diabetes mellitus or signs of organ failure (anaemia, kidney failure, liver failure, etc)
* misuse/dependency of alcohol, sedatives, neurostimulating or narcotic drugs)
* obstructive sleep apnoea/hypopnoea syndrome
* using CPAP/BiPAP or home respirator
* pregnancy
* if PSG shows AHI > 30, or if patient becomes acutely ill between the nights with PSG, he/she will be withdrawn from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
transcutaneously measured pCO2 during sleep | 1 year

SECONDARY OUTCOMES:
cardiac arrythmias registered by Holter monitoring | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nils H Holmedahl, MD, Principal Investigator — LHL Helse
Locations (2):
- Norway (2):
  - Glittreklinikken, Hakadal, Akershus
  - Glittreklinikken, Oslo, Hakadal